CLINICAL TRIAL: NCT06566859
Title: Comparison of ESP Block and M-TAPA Block Efficiency in Postoperative Analgesia Management in Nephrectomy Cases
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Hilal AKCA, MD, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024-297
Record Dates: First submitted 2024-08-11; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative
Keywords: nerve block; pain management; postoperative period; postoperative complications; regional anesthesia; pain
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Postoperative Complications; Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- M-TAPA Block: Patients who have standard anesthesia are randomized with the research randomizer application while under anesthesia and M-TAPA block is applied under ultrasound guidance in the preoperative period. For the block, 50 mg of 0.25% bupivacaine and 100 mg lidocaine are injected, totaling 20cc.
  Interventions: Other: NRS 0. hour; Other: NRS 6. Hour; Other: NRS 12. Hour; Other: NRS 24. Hour
- ESP Block: Patients who have standard anesthesia are randomized with the research randomizer application while under anesthesia and ESP block is applied under ultrasound guidance in the preoperative period. For the block, 50 mg of 0.25% bupivacaine and 100 mg lidocaine are injected, totaling 20cc.
  Interventions: Other: NRS 0. hour; Other: NRS 6. Hour; Other: NRS 12. Hour; Other: NRS 24. Hour

INTERVENTIONS:
Other: NRS 0. hour — Numerical rating scala
Other: NRS 6. Hour — Numerical rating scala
Other: NRS 12. Hour — Numerical rating scala
Other: NRS 24. Hour — Numerical rating scala

SUMMARY:
Relieving postoperative nephrectomy pain requires multimodal approaches. Peripheral blocks such as ESP block and M-TAPA block and multimodal analgesics reduce side effects by reducing the use of other analgesics. This study aimed to compare the effectiveness of erector spinae plane block (ESP block) and modified thoracoabdominal nerve blocking with perichondrial approach (M-TAPA block) in postoperative analgesia management in nephrectomy cases.

DETAILED DESCRIPTION:
Relieving postoperative nephrectomy pain requires multimodal approaches. The most commonly used in the treatment of pain are nonsteroidal anti-inflammatory drugs (NSAIDs), opioids, and infiltration of local anesthetics. Due to the side effects of NSAIDs and opioids, the application of regional analgesia techniques can reduce complications while providing better analgesia quality. Peripheral blocks such as ESP block and M-TAPA block and multimodal analgesics reduce side effects by reducing the use of other analgesics. Pain is considered one of the most important factors affecting the quality of healing. Postoperative pain delays the postanesthesia care unit, hospital stay, early ambulation, increases resource utilization, and negatively affects patient satisfaction. If postoperative analgesia is provided, all these negativities will be eliminated. This study aimed to compare the effectiveness of erector spinae plane block (ESP block) and modified thoracoabdominal nerve blocking with perichondrial approach (M-TAPA block) in postoperative analgesia management in nephrectomy cases.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and over with ASA1-2 who underwent elective nephrectomy

Exclusion Criteria:

* ASA ≥3
* Body mass index>35 kg/ m²
* Infection in the block area
* Coagulation disorder,
* Known allergy to local anesthetics
* Pregnant
* Patient with neuropathy
* Patient without cooperation
* Patient who refuses to participate in the study
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 and over with ASA1-2 who underwent elective nephrectomy.
  .
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Management | 0.hour
  The primary outcome of this study is to demonstrate that Modified Thoracoabdominal Nerves Block(M-TAPA) contributes sufficiently to multimodal analgesia in perioperative analgesia in nephrectomy surgery.This contribution will be evaluated with the NRS. NRS is a unidimensional scale in which 11 numbers (between 0 and 10) are used to measure pain intensity. The patient is asked to choose the number that best reflects the pain intensity, with 0 = no pain and 10 = worst (unbearable) pain.
Postoperative Pain Management | 6.hour
  The primary outcome of this study is to demonstrate that Modified Thoracoabdominal Nerves Block(M-TAPA) contributes sufficiently to multimodal analgesia in perioperative analgesia in nephrectomy surgery.This contribution will be evaluated with the NRS. NRS is a unidimensional scale in which 11 numbers (between 0 and 10) are used to measure pain intensity. The patient is asked to choose the number that best reflects the pain intensity, with 0 = no pain and 10 = worst (unbearable) pain.
Postoperative Pain Management | 12.hour
  The primary outcome of this study is to demonstrate that Modified Thoracoabdominal Nerves Block(M-TAPA) contributes sufficiently to multimodal analgesia in perioperative analgesia in nephrectomy surgery.This contribution will be evaluated with the NRS. NRS is a unidimensional scale in which 11 numbers (between 0 and 10) are used to measure pain intensity. The patient is asked to choose the number that best reflects the pain intensity, with 0 = no pain and 10 = worst (unbearable) pain.
Postoperative Pain Management | 24.hour
  The primary outcome of this study is to demonstrate that Modified Thoracoabdominal Nerves Block(M-TAPA) contributes sufficiently to multimodal analgesia in perioperative analgesia in nephrectomy surgery.This contribution will be evaluated with the NRS. NRS is a unidimensional scale in which 11 numbers (between 0 and 10) are used to measure pain intensity. The patient is asked to choose the number that best reflects the pain intensity, with 0 = no pain and 10 = worst (unbearable) pain.
Postoperative Pain Management | 24 hours
  Total amount of analgesic used in 24 hours
Postoperative Pain Management | 24 hours
  Time of first additional analgesic requirement up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Akça, Principal Investigator — BasaksehirCamSakuraH
Locations (1):
- BasaksehirCamSakuraH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided